CLINICAL TRIAL: NCT03079323
Title: Phase II Trial to Investigate the Benefit of Elective Para-Aortic Radiotherapy (PART) for pN1 Prostate Cancer Using Arc Therapy (IMAT/VMAT)
Brief Title: Trial to Investigate the Benefit of Elective Para-Aortic Radiotherapy (PART) for pN1 Prostate Cancer
Acronym: PART
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S59533
Record Dates: First submitted 2017-02-23; First posted 2017-03-14 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer
Keywords: External beam radiotherapy; Prostate cancer; Elective para-aortic radiation therapy; PART
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PART-trial (Experimental): External beam radiotherapy
  Interventions: Radiation: PART-trial

INTERVENTIONS:
Radiation: PART-trial — Elective radiation to the para-aortic lymph nodes 45 Gy / 1.8 Gy

SUMMARY:
Prospective non-randomized phase 2 trial to study the efficacy of additional elective para-aortic RT (PART) in pN1 patients compared to those who were historically treated with adjuvant whole pelvic radiotherapy (WPRT) alone.

DETAILED DESCRIPTION:
Rationale: In prostate cancer with histopathologically proven pelvic lymph node metastasis (pN1) after extended pelvic lymph node dissection, multimodality treatment consisting of treatment of the primary tumor, androgen deprivation therapy and whole pelvic radiotherapy offers the best results and is the standard-of-care. However, in case >1 pelvic lymph node is invaded by tumor, after extended pelvic lymph node dissection, 40% of the patients relapse biochemically and clinically. Clinical relapse is present in the para-aortic lymph nodes (M1a disease) in 25% of the cases as we observed in series. Therefore Elective Para-Aortic Radiotherapy (PART) may improve disease control.

Objective: The main goal of this phase II study is to investigate whether elective para-aortic radiotherapy increases the clinical relapse-free survival (cRFS) defined as the absence of clinical relapse (cR) at biological imaging at 5 years. The secondary objectives of this study are: acute toxicity, late toxicity, quality of life (QoL), time to palliative androgen deprivation therapy (ADT), time to castration refractory prostate cancer (CRPC), cause-specific survival and in field pelvic and para-aortic disease control.

Study design: The PART-trial is a non-randomized phase II trial.

Study population: Men with histological proven adenocarcinoma of the prostate (cT1-4; pT2-4) and presence of pN1 disease after ePLND are eligible for the study. For trial-inclusion, pN1 disease is defined on the basis of one of following criteria: (1) two or more positive LN; (2) ratio positive LN / removed LN > 7%; (3) presence of extracapsular LN extension. Patients referred for external beam radiotherapy (EBRT) who fulfill the inclusion criteria and without any of the exclusion criteria will be included in the present trial after written informed consent.

Intervention: Patients included in the PART-trial receive radiotherapy to the prostate or prostate bed and the pelvic lymph nodes according to the current standard. Furthermore patients in the PART-trial receive an additional elective radiation to the para-aortic lymph nodes. The total radiation dose that will be delivered to the para-aortic lymph node area is 45 Gy in 25 fractions of 1.8 Gy. Androgen deprivation therapy is foreseen in this trial for 24 months (long term).

Main study parameters/endpoints: The primary endpoint is to evaluate whether the addition of an elective para-aortic irradiation for pN1 prostate cancer patients increases the clinical relapse-free survival (cRFS) defined as the absence of clinical relapse (cR) at biological imaging at 5 years. Clinical relapse-free survival is defined by a combination of PSA measurements and imaging. Secondary endpoints are acute and late gastrointestinal (GI) and genitourinary (GU) toxicity using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, QoL, time to palliative ADT, time to CRPC, cause-specific survival and in field pelvic and para-aortic disease control.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and willingness to comply with the treatment and follow-up
* Diagnosis of histopathologically confirmed prostate cancer
* No former treatment for prostate cancer
* Presence of pN1 disease after ePLND (criteria defined in the protocol)
* Age > 18
* Karnofsky Performance score > 70
* Ability to understand the informed consent (Helsinki Declaration)

Exclusion Criteria:

* Recurrent disease status
* Presence of cM1a, cM1b or cM1c disease
* Former radiotherapy making WPRT and/or PART impossible
* Prior malignancy, not disease-free > 5 years, except basocellular skin epithelioma
* Severe or active comorbidity likely to impact on the feasibility of WPRT and/or PART
* Disorder precluding understanding of trial information

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2017-02-06 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Clinical relapse-free survival (cRFS) | Median follow-up of 60 months
  The absence of clinical relapse (cR) at biological imaging

SECONDARY OUTCOMES:
Acute toxicity | Median follow-up of 90 days
  (CTCAE 4.0)
Late toxicity | Median follow-up of 3 years
  (CTCAE 4.0)
Quality-of-life - General | Median follow-up of 3 years
  EORTC QLQ-C30
Quality-of-life - Prostate specific | Median follow-up of 3 years
  EORTC QLQ-PR25
Quality-of-life - Measure of health outcome | Median follow-up of 3 years
  EQ-5D-5L
Quality-of-life - Urinary incontinence | Median follow-up of 3 years
  ICIQ-SF
Quality-of-life - Erectile function | Median follow-up of 3 years
  IIEF-5
Time to palliative ADT | Median follow-up of 5 years
  Indications for palliative ADT or based on the EAU guidelines
Time to castration-refractory prostate cancer (CRPC) | Median follow-up of 5 years
  Criteria for CRPC as defined in the EAU guidelines
Cause-specific survival | Median follow-up of 5 years
  Cause-specific survival
Overall survival | Median follow-up of 5 years
  Overall survival
In field pelvic disease control (at biological imaging) | Median follow-up of 5 years
  In field pelvic disease control (PET-CT imaging (PSMA/choline) is performed in case of PSA progression)
In field PA disease control (at biological imaging) | Median follow-up of 5 years
  In field PA disease control (PET-CT imaging (PSMA/choline) is performed in case of PSA progression)

CONTACTS AND LOCATIONS:
Overall Officials: Gert De Meerleer, Prof. Dr., Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Draulans C, Joniau S, Fonteyne V, Delrue L, Decaestecker K, Everaerts W, Dirix P, Van den Bergh L, Crijns W, Vandendriessche H, Van Wynsberge L, Ost P, Lumen N, Buelens P, Haustermans K, Berghen C, De Meerleer G. Benefits of Elective Para-Aortic Radiotherapy for pN1 Prostate Cancer Using Arc Therapy (Intensity-Modulated or Volumetric Modulated Arc Therapy): Protocol for a Nonrandomized Phase II Trial. JMIR Res Protoc. 2018 Dec 13;7(12):e11256. doi: 10.2196/11256. PMID 30545809